CLINICAL TRIAL: NCT01119742
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Design, Multiple-Site Study to Evaluate the Clinical Equivalence of Two Generic Butenafine Hydrochloride 1% Creams to Lotrimin Ultra® Cream in Patients With Interdigital Tinea Pedis
Brief Title: Clinical Equivalence of Two Generic Butenafine Hydrochloride 1% Creams as Compared to Lotrimin Ultra Cream in Patients With Interdigital Tinea Pedis
Acronym: BNF-0909
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient number of baseline eligible patient
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTNF-0909
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Interdigital Tinea Pedis
Keywords: Tinea Pedis; Interdigital
MeSH Terms: conditions — Tinea Pedis | interventions — butenafine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Butenafine Hydrochloride 1% A (Experimental): 1
  Interventions: Drug: Butenafine Hydrochloride 1%
- Butenafine Hydrochloride 1% B (Experimental): 2
  Interventions: Drug: Butenafine Hydrochloride 1% B
- Butenafine Hydrochloride 1% (Active Comparator): 3
  Interventions: Drug: Butenafine Hydrochloride 1%
- Vehicle A (Placebo Comparator): 4
  Interventions: Drug: Vehicle A
- Vehicle B (Placebo Comparator): 5
  Interventions: Drug: Vehicle B

INTERVENTIONS:
Drug: Butenafine Hydrochloride 1% — Twice daily application for 7 days
  Arms: Butenafine Hydrochloride 1% A
Drug: Butenafine Hydrochloride 1% B — Twice daily application for 7 days
  Arms: Butenafine Hydrochloride 1% B
Drug: Butenafine Hydrochloride 1% — Twice daily application for 7 days
  Other Names: Lotrimin Ultra Cream
  Arms: Butenafine Hydrochloride 1%
Drug: Vehicle A — Twice daily application for 7 days
  Arms: Vehicle A
Drug: Vehicle B — Twice daily application for 7 days
  Arms: Vehicle B

SUMMARY:
To demonstrate comparable safety and efficacy of Taro Pharmaceuticals, Inc butenafine hydrochloride cream 1% test product and Lotrimin Ultra cream (reference listed drug) in the treatment of interdigital tinea pedis, and to show the superiority of the active treatments over that of the placebo (vehicle).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non lactating females 18 years of age or older.
2. Signed informed consent form, which meets all criteria of current FDA regulations and the requirements of the India regulatory authorities.
3. If female and of child bearing potential, have a negative urine pregnancy test at the baseline visit,
4. A total score of at least six (6) for the following eight (8) clinical signs and symptoms of interdigital tinea pedis: fissuring, erythema, maceration, vesiculation, desquamation/scaling, exudation, pruritus, burning/stinging. In addition the most infected area must have a minimum score of at least 2 for erythema and a minimum score of at least 2 for either pruritus or desquamation/scaling
5. A confirmed clinical diagnosis of interdigital tinea pedis.
6. The presence of tinea pedis infection, confirmed by the observation of segmented fungal hyphae during a microscopic KOH wet mount examination (potassium hydroxide mount preparation).
7. Identification of an appropriate dermatophyte by culture sent to the central laboratory. The appropriate dermatophytes are Trichophyton rubrum, Trichophyton mentagrophytes or Epidermophyton floccosum.

Exclusion Criteria:

1. Use of any of the following within the indicated timeline:

   * Oral or injectable steroids within four weeks of the study start.
   * Any oral anti-fungals within 4 weeks of the study start.
   * Use of topical corticosteroids or any other topical antipruritics on the feet within 72 hours of the study start.
   * Any prescription or OTC topical antifungal on the feet within two weeks prior to study entry.
   * Use of any antihistamines within 72 hours of the study start.
2. Any known hypersensitivity to butenafine or other antifungal agents.
3. Evidence of any concurrent dermatophytic infection of toe nails (onychomycosis) or other dermatological condition of the foot that may interfere with the Investigators evaluation of tinea pedis.
4. Patients with recurrent tinea pedis (more than 3 infections in the past 12 months) who have been unresponsive to previous antifungal therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure | 42 Days
  Patients with clinical cure and mycologic cure are considered therapeutic cures.

SECONDARY OUTCOMES:
Clinical Cure | 42 days
  Patient will be considered a "clincal cure" if the score for erythema is equal or less than 2 and the total score for all of the other seven signs and symptoms is less than 2.
Mycologic Cure | 42 Days
  Patient will be considered a "mycological cure" if the results of both the potassium hydroxide (KOH) and the fungal culture are negative.